CLINICAL TRIAL: NCT05780944
Title: Does Paced Bottle-Feeding Improve the Quality and Outcome of Bottle-Feeding Interactions?
Brief Title: Short-term Effects of Paced Bottle-Feeding on Feeding Interactions
Acronym: PBF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Responsible Party: Principal Investigator, Alison Ventura, Associate Professor, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-253-CP
Record Dates: First submitted 2023-02-28; First posted 2023-03-23 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Mother-Infant Interaction; Breastfeeding; Bottle Feeding
Keywords: paced bottle-feeding; feeding interactions; maternal feeding practices; responsive feeding; infant feeding; breastfeeding; bottle-feeding
MeSH Terms: conditions — Breast Feeding; Bottle Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: After each visit, three trained coders who are unaware of the experimental conditions and hypotheses of the study will score the videotaped records using an event recorder program (Observer XT, version 16; Noldus Information Technology, Heerlen, the Netherlands).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding First, Bottle-feeding Second, PBF Third (Experimental): Mother-infant dyads will visit the laboratory on three different days. During the first visit, they will be observed during breastfeeding. During the second visit, they will be observed during bottle-feeding. During the third visit, the mother will be taught the PBF approach and will be observed using it during bottle-feeding.
  Interventions: Behavioral: Paced Bottle-Feeding Education
- Bottle-feeding First, Breastfeeding Second, PBF Third (Experimental): Mother-infant dyads will visit the laboratory on three different days. During the first visit, they will be observed during bottle-feeding. During the second visit, they will be observed during breastfeeding. During the third visit, the mother will be taught the PBF approach and will be observed using it during bottle-feeding.
  Interventions: Behavioral: Paced Bottle-Feeding Education

INTERVENTIONS:
Behavioral: Paced Bottle-Feeding Education — Participants will be asked to review an educational handout that outlines how to implement PBF during bottle-feeding interactions. Participants will then be asked to watch a video that further describes PBF and illustrates how to implement it with a live infant. A trained research assistant will then answer questions, further explain PBF, and demonstrate PBF with a baby doll, using a standardized script

SUMMARY:
Current infant feeding recommendations focus on promoting responsive feeding, which is widely recognized as the ideal way to feed infants because it is associated with healthier eating behaviors and growth outcomes for infants. Unfortunately, many bottle-feeding families receive inadequate support for learning responsive bottle-feeding practices because breastfeeding support is prioritized in healthcare settings. Promotion of breastfeeding is an important focus for public health efforts, but a significant proportion of families bottle-feed their infants, either exclusively or in combination with breastfeeding. Thus, bottle-feeding remains a ubiquitous part of infant feeding and evidence-based strategies are needed to support bottle-feeding families. One promising strategy is the Paced Bottle-Feeding (PBF) method, which incorporates many ideas and feeding practices consistent with the concept of responsive feeding. This approach to bottle-feeding aims to mimic the aspects of breastfeeding that promote balanced control between caregiver and infant and allow the infant to set the pace of the feeding in response to feelings of hunger and fullness. Although PBF is sometimes taught in perinatal education settings, teaching new parents about PBF is not an evidence-based practice because there have been no empirical studies evaluating the effectiveness of PBF for promoting responsive feeding for parents and healthy intake and weight outcomes for infants. Thus, despite the conceptual promise of PBF for promoting responsive bottle-feeding interactions, research is needed to determine whether PBF is effective and identify whether any limitations of this method exist. This study is a within-subject, experimental study wherein mother-infant dyads will be observed during breastfeeding and typical bottle-feeding interactions. Mothers will then be taught the PBF method and observed during a PBF interaction. This design will allow for direct testing of the purported benefits of PBF over typical bottle-feeding and whether PBF makes the experience of bottle-feeding more equivalent to the experience of breastfeeding. The overarching aims of this study are to explore the ways in which bottle-feeding can go well and identify mechanisms through which bottle-feeding families can be supported to promote healthy intake and weight gain trajectories for their infants.

DETAILED DESCRIPTION:
Infancy is a sensitive period for obesity prevention efforts, in part because rapid weight gain during infancy is a stronger predictor of later obesity and metabolic comorbidities than weight gain trajectories during later life. The first 6 months are of particular importance given research illustrating overfeeding during this early window places infants at significantly higher risk for rapid weight gain compared to overfeeding during later infancy. To prevent overfeeding and rapid weight gain, current recommendations and prevention programs primarily focus on promoting responsive feeding during infant feeding interactions.

During responsive feeding, infants are fed in ways that are developmentally appropriate and responsive to infant hunger and fullness cues. Responsive feeding is widely recognized as the ideal way to feed infants because it gives them the scaffolded support to learn to recognize and eat in response to hunger and fullness cues and to self-regulate intake in response to physiological needs. Indeed, responsive feeding is associated with healthier eating behaviors and growth outcomes for infants.

Promotion of responsive feeding is typically a core component of breastfeeding promotion and education. However, a significant proportion of families bottle-feed their infants, either exclusively or in combination with breastfeeding. U.S. data illustrate 42% of infants are exclusively bottle-fed by 6 months of age and 70% of breastfed infants receive supplemental formula or bottle-feedings on a regular basis. Thus, bottle-feeding is a ubiquitous part of infant feeding and evidence-based strategies are needed to complement breastfeeding education and promote responsive bottle-feeding.

Unfortunately, many bottle-feeding families receive inadequate support for learning responsive bottle-feeding, likely because breastfeeding support is prioritized in health care settings. In addition, mothers perceive health professionals to be ill-prepared to help them with their formula- and bottle-feeding needs and reluctant to discuss formula- or bottle-feeding at the risk of compromising breastfeeding support. A striking 1 in 5 formula-feeding mothers reported they received no advice related to infant feeding from health care professionals compared to only 5% of breastfeeding mothers.

To date, few studies address this need, creating a significant research gap that hinders support for bottle-feeding families. Thus, promotion of responsive bottle-feeding remains a realistic but under-utilized facet of early support. One promising strategy is the "paced-bottle feeding" (PBF) method, which incorporates many concepts and strategies consistent with the concept of responsive feeding.

PBF was first introduced by a lactation consultant to reduce nipple confusion and bottle-preference among breastfeeding infants being introduced to bottles. In brief, to implement PBF, caregivers are taught to:

* Initiate feeding when the infant shows hunger cues (e.g., rooting, sucking noises).
* Hold the infant during the entire feeding and avoid propping the bottle on a blanket or leaving the feeding infant unattended.
* Hold the bottle horizontal so that the nipple is only partially full of milk and hold the infant upright instead of a more prone position to moderate milk flow and encourage the infant to actively work to remove milk.
* When offering the bottle, allow the infant to take the nipple rather than pushing or forcing the nipple into the infant's mouth
* Allow the infant to pause and take breaks
* Switch the infant from one side to the other during the feeding (just like a mother would switch breasts)
* Allow at least 15-20 minutes for feeding so the infant has enough time to feel full
* Terminate feeding when the infant exhibits fullness cues (e.g., slowing pace of feeding, turning away); refrain from encouraging the infant to finish the bottle

The purported (but untested) benefits of PBF stem from the idea that PBF makes the experience of bottle-feeding more equivalent to the experience of breastfeeding by slowing the pace of feeding and increasing the amount of effort infants expend during bottle-feeding. Proponents of PBF claim that these features of PBF promote balanced control between caregiver and infant wherein the infant is better able to set the pace of feeding and stop feeding when full, reducing risk for spitting up and overfeeding.

Since its introduction in 2002, education about PBF during prenatal breastfeeding classes has grown in popularity. Additionally, the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) began to incorporate PBF into their infant feeding education curriculum for both breast- and formula-feeding mothers. Although promising, teaching new parents PBF is not an evidence-based practice because there have been no empirical studies evaluating the effectiveness of PBF for promoting responsive feeding and healthy intake and weight outcomes for infants. Thus, despite the conceptual promise of PBF for promoting responsive bottle-feeding, research is needed to determine whether PBF is effective and observe whether any limitations of the method exist.

The objective of this project will be to address this research gap by comparing short-term feeding interactions and outcomes during PBF to both breastfeeding and typical bottle-feeding. This study is a within-subject experimental study of 60 mother-infant dyads who are both breast- and bottle-feeding. Within this study, mothers will be observed during breastfeeding and typical bottle-feeding interactions. Mothers will then be taught the PBF method and observed during a PBF interaction.

This study will address the following specific aims:

Aim 1: To test the hypothesis that PBF will lead to significantly lower infant milk intake (mL), longer meal duration (min), slower rate of feeding (mL/min), and lower frequency of spitting up compared to typical bottle-feeding, but similar intake, meal duration, rate of feeding, and frequency spitting up compared to breastfeeding.

Aim 2: To test the hypothesis that mothers will exhibit greater sensitivity and responsiveness to infant cues during PBF compared to typical bottle-feeding, but similar sensitivity and responsiveness to infant cues compared to breastfeeding.

Aim 3: To test the hypothesis that infants will exhibit greater clarity of cues and responsiveness to feeding during PBF compared to typical bottle-feeding, but similar clarity of cues and responsiveness to feeding compared to breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Speaks English or Spanish
* Mother 18-40-years of age
* Infant 0-24 weeks of age
* Dyad is current breastfeeding and bottle-feeding
* Infant has not been introduced to solid foods

Exclusion Criteria:

* Infant was born preterm (<37 weeks)

Max Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Infant Milk Intake between Breastfeeding, Typical Bottle-Feeding, and Paced Bottle-Feeding Conditions | 3 visits across a 1 week period
  Infant milk intake in mL, assessed by weighing the infant before and after each feeding condition
Change in Meal Duration between Breastfeeding, Typical Bottle-Feeding, and Paced Bottle-Feeding Conditions | 3 visits across a 1 week period
  Duration of the observed meal in minutes (min), determined by trained video coders masked to study hypotheses
Change in Rate of Feeding between Breastfeeding, Typical Bottle-Feeding, and Paced Bottle-Feeding Conditions | 3 visits across a 1 week period
  Infant milk intake divided by meal duration (mL/min)
Change in Frequency of Spitting Up During and After the Meal between Breastfeeding, Typical Bottle-Feeding, and Paced Bottle-Feeding Conditions | 3 visits across a 1 week period
  Determined by trained video coders masked to study hypotheses
Change in Maternal Sensitivity to Infant Cues between Breastfeeding, Typical Bottle-Feeding, and Paced Bottle-Feeding Conditions | 3 visits across a 1 week period
  Determined by video coders masked to study hypotheses and certified in the Nursing Child Assessment Caregiver-Child Interaction Feeding Scale (NCAFS); possible Maternal Sensitivity to Infant Cues scores range from 0-16 with higher scores representing greater maternal sensitivity to infant cues
Change in Maternal Responsiveness to Infant Distress between Breastfeeding, Typical Bottle-Feeding, and Paced Bottle-Feeding Conditions | 3 visits across a 1 week period
  Determined by video coders masked to study hypotheses and certified in the Nursing Child Assessment Caregiver-Child Interaction Feeding Scale (NCAFS); possible Maternal Responsiveness to Infant Distress scores range from 0-11 with higher scores representing greater maternal responsiveness to infant distress
Change in Infant Clarity of Cues between Breastfeeding, Typical Bottle-Feeding, and Paced Bottle-Feeding Conditions | 3 visits across a 1 week period
  Determined by video coders masked to study hypotheses and certified in the Nursing Child Assessment Caregiver-Child Interaction Feeding Scale (NCAFS); possible Infant Clarity of Cues scores range from 0-15 with higher scores representing greater infant clarity of cues
Change in Infant Responsiveness to Caregiver between Breastfeeding, Typical Bottle-Feeding, and Paced Bottle-Feeding Conditions | 3 visits across a 1 week period
  Determined by video coders masked to study hypotheses and certified in the Nursing Child Assessment Caregiver-Child Interaction Feeding Scale (NCAFS); possible Infant Responsiveness to Caregiver scores range from 0-11 with higher scores representing greater infant responsiveness to the caregiver

CONTACTS AND LOCATIONS:
Overall Officials: Alison K Ventura, PhD, Principal Investigator — Associate Professor
Locations (1):
- California Polytechnic State University, San Luis Obispo, California, United States

IPD SHARING:
Plan to Share IPD: No
The research team is willing to share deidentified data with other researchers. Interested researchers can contract the principal investigator to request access to the data.

REFERENCES:
- See also: Study Website — https://healthykids.calpoly.edu/pacedbottlefeeding